CLINICAL TRIAL: NCT03988673
Title: Comparison of Explicit Values Clarification Method (VCM), Implicit VCM and no VCM Decision Aids for Men Considering Prostate Cancer Screening: Protocol of a Randomized Trial
Brief Title: Comparison of Explicit, Implicit and no Values Clarification Decision Aids for Men Considering Prostate Cancer Screening
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Universidade do Porto (Other)
Collaborators: NOVA Medical School (Other); Georgetown University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Other
Other Study IDs: DA-VCM
Record Dates: First submitted 2019-06-03; First posted 2019-06-17 (Actual); Last update posted 2019-06-17 (Actual); Status verified 2019-05

CONDITIONS: Healthy Volunteers
MeSH Terms: interventions — Decision Support Techniques

STUDY DESIGN:
Intervention Model Description: Parallel three group (1:1:1): (i) decision aid with information only (Control), (ii) decision aid with information plus an implicit VCM, (iii) decision aid with information plus an explicit VCM.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- decision aid with information only (control) (No Intervention): decision aid with information only, without values clarification method (VCM)
- decision aid with implicit VCM (Active Comparator): decision aid with information plus an implicit VCM
  Interventions: Other: Decision aid with implicit values clarification method (booklet or website)
- decision aid with explicit VCM (Active Comparator): decision aid with information plus an explicit VCM
  Interventions: Other: Decision aid with explicit values clarification method (booklet or website)

INTERVENTIONS:
Other: Decision aid with implicit values clarification method (booklet or website) — The intervention will be an informative evidence-based material in the format of a booklet or website concerning prostate cancer screening. The values clarification method will be a grid where statements about the subject will be presented (decision aid with implicit VCM).
  Arms: decision aid with implicit VCM
Other: Decision aid with explicit values clarification method (booklet or website) — The intervention will be an informative evidence-based material in the format of a booklet or website concerning prostate cancer screening. The values clarification method will be a a grid where statements about the subject will be presented and men should indicate what statements they identify with (decision aid with explicit VCM).
  Arms: decision aid with explicit VCM

SUMMARY:
The investigators aim at comparing the perceived clarity of personal values in men considering PSA screening using decision aids with no VCM versus an implicit VCM versus an explicit VCM. This study will add to the body of evidence on the role of decision aids to support health preference-sensitive choices and provide further insight on the impact of different methods for eliciting people's values embedded within a decision aid.

DETAILED DESCRIPTION:
PSA test to screen for prostate cancer is considered a preference sensitive decision, meaning it does not only depend on what is best from a medical point of view, but also on patient values. Decision aids are evidence-based tools which showed to help people feel clearer about their values, therefore it has been advocated that decision aids should contain a specific values clarification method (VCM). VCM may be either implicit or explicit but the evidence concerning the best method is scarce. We aim at comparing the perceived clarity of personal values in men considering PSA screening using decision aids with no VCM versus an implicit VCM versus an explicit VCM.

ELIGIBILITY:
Inclusion Criteria:

* adult men (50 - 69 years);
* men with average risk for prostate cancer;
* willing and able to provide written informed consent.

Exclusion Criteria:

* unable to understand written Portuguese.

Ages: 50 Years to 69 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Gender Based: Yes — the intervention's purpose is to support men's prostate cancer screening decision
Enrollment: 276 (Estimated)
Dates: Start 2019-09 (Estimated); Primary Completion 2019-12 (Estimated); Study Completion 2020-09 (Estimated)

PRIMARY OUTCOMES:
Perceived clarity of personal values | immediately after the intervention
  3-item subscale of the Decisional Conflict Scale. Items are given a score of 0 ("strongly agree") to 4 ("strongly disagree"). Items are: a) summed; b) divided 3; and c) multiplied by 25. Scores range from 0 [feels extremely clear about personal values] to 100 [feels extremely unclear about personal values].

SECONDARY OUTCOMES:
Decisional Conflict | immediately after the intervention
  Decisional Conflict Scale (16-item). Items are given a score of 0 ("strongly agree") to 4 ("strongly disagree"). Items are: a) summed; b) divided 16; and c) multiplied by 25. Scores range from 0 [no decisional conflict] to 100 [extremely high decisional conflict].
% of patients with preference to undergo PSA screening (screening intention; questionnaire) | before and immediately after the intervention
  Intention to undergo prostate cancer screening with PSA: questionnaire - single question about intention to be screened with PSA, using a 5 point-Likert scale (ranging from "strongly disagree" to "strongly agree"; intention to undergo PSA screening will be considered positive if the respondent replies with "agree" or "strongly agree"). % of patients with preference to undergo PSA screening.
% of patients who underwent PSA screening (questionnaire) | 6 months after the intervention
  Self-reported PSA screening. Questionnaire - single question. Men will report wether they have or have not underwent PSA screening after the intervention. % of patients who underwent PSA screening

CONTACTS AND LOCATIONS:
Overall Officials: Sofia Baptista, MD, Principal Investigator — Universidade do Porto

IPD SHARING:
Plan to Share IPD: No
Data will be made available on request

REFERENCES:
- [Derived] Baptista S, Heleno B, Teixeira A, Taylor KL, Martins C. Comparison of explicit values clarification method (VCM), implicit VCM and no VCM decision aids for men considering prostate cancer screening: protocol of a randomized trial. BMC Med Inform Decis Mak. 2020 Apr 29;20(1):78. doi: 10.1186/s12911-020-1094-3. PMID 32349746